CLINICAL TRIAL: NCT03750422
Title: A Split-body, Double-blinded, Placebo-controlled Trial of Stratacel® Wound Dressing After Laser Treatment of Striae Alba
Brief Title: Stretch Marks on Abdomen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Principal Investigator, Isabella Guiha, CCRC, Goldman, Butterwick, Fitzpatrick and Groff
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STRATPHARMA-2018-01
Record Dates: First submitted 2018-11-08; First posted 2018-11-23 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Striae; Albicantes
MeSH Terms: conditions — Striae Distensae | interventions — Aquasonic

STUDY DESIGN:
Intervention Model Description: double-blinded, randomized split-body study
Who Masked: Participant, Investigator
Masking Description: Subjects are provided with de-identified tubes of both study product and vehicle then instructed on which de-identified product is to be used for aftercare on which side of the abdomen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Stratacel (Active Comparator): medical grade silicone gel following Picoway Laser treatment
  Interventions: Device: Picoway; Other: Stratacel
- Vehicle (Sham Comparator): Clear ultrasound gel following Picoway Laser treatment
  Interventions: Device: Picoway; Other: Aquasonic

INTERVENTIONS:
Device: Picoway — 1064/532nm picosecond laser
Other: Stratacel — a self-drying, bacteriostatic, transparent silicone gel with anti-inflammatory properties
  Arms: Stratacel
Other: Aquasonic — clear ultrasound gel
  Arms: Vehicle

SUMMARY:
The primary objective of this study is to determine the effect of Stratacel® wound dressing on cosmetic outcomes following 1064/532nm picosecond laser (Picoway®, Syneron Candela Corp, Wayland, MA, USA) treatment of abdominal striae alba. Secondary objectives include examining the effect of Stratacel® wound dressing on post-laser healing and symptomatology.

DETAILED DESCRIPTION:
Twenty adult subjects with abdominal striae alba will be enrolled. All striae will be treated using the 1064/532nm picosecond laser with designated and standardized settings (Appendix A). The abdominal striae treatment region will then be split across the body vertically with one half randomized to Stratacel® and the other to placebo, clear ultrasound gel (Aquasonic). A blinded study coordinator will apply the products to each randomized half-abdomen immediately following laser treatment.

A total of 3 treatments will be completed at 1 month intervals. Blinded-investigator and subject self-assessments will be performed at post-treatment days 2, 5, 7, and 10 after each laser session. Assessments will also be performed 1 and 3 months after the final laser treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Females or Males in good general health >18 years of age.
2. Must be willing to give and sign a photography release, HIPPA and informed consent.
3. Subject must have at least 2 white striae on each treatment side of the abdomen that measure at least 1cm in length.
4. Females will be either of non-childbearing potential defined as:

1. Having no uterus 2. No menses for at least 12 months.

Or:

Women of childbearing potential must agree to use an effective method of birth control during the course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment participation. Expectable forms of birth control below:

1. Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device
2. Intrauterine coil
3. Bilateral tubal ligation
4. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
5. Abstinence (If practicing abstinence must agree to use barrier method described above (4) if becomes sexually active).
6. Vasectomized (must agree to use barrier method described above (4) if becomes sexually active with un-vasectomized partner).

Exclusion Criteria:

1. Pregnancy, planned pregnancy during the course of the study or currently breast feeding.

2. Projected significant fluctuations in weight during the course of the study or within the last 6 months, per investigator discretion.

1. Recent use of self-tanners, excessive exposure to sunlight, artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing) or expectations of tanning and/or use of self-tanners during the course of the study.
2. Any planned surgical or cosmetic procedure in the treatment area during the course of the study.
3. Any UNCONTROLLED systemic disease -a potential patient in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study.
4. Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
5. Red or brown colored striae in the intended treatment area.
6. Active dermatitis, open wound, active bacterial, neurologic, fungal, or viral infection in the proposed treatment area.
7. Inability to ambulate following the procedure.
8. History of skin tightening or other treatment in the striae region in the preceding 12 months before study enrollment and for duration of the study.
9. Use of topical retinoids, hydroquinone, medicated cleansers, cellulite creams, or steroids to the treatment area within the preceding 2 weeks and for duration of the study.
10. Allergy to any ingredient in the study medication or placebo.
11. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Striae Texture | Pre-Treatment to 3-months post final treatment.
  Assessment of texture Pre treatment and post final treatment using a 5-Point Blinded Investigator Striae Assessment scale
Change in Striae Color | Pre-Treatment to 3-months post final treatment.
  Assessment of Color Pre treatment and post final treatment
Change in Striae Size | Pre-Treatment to 3-months post final treatment.
  Assessment of Size Pre treatment and post final treatment using a 5-Point Blinded Investigator Striae Assessment scale.
Change in Striae Overall Appearance | Pre-Treatment to 3-months post final treatment.
  Assessment of Overall Appearance Pre treatment and post final treatment using a 6-Point Blinded Investigator Striae Assessment scale

SECONDARY OUTCOMES:
Safety - Post Laser Treatment Adverse Events | days 2, 5, 7, and 10 after each laser session
  erythema, edema, crusting, bruising, hyperpigmentation, hypopigmentation, and scarring

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — Cosmetic Laser Dermatology
Locations (1):
- West Dermatology Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No